CLINICAL TRIAL: NCT01135108
Title: A Double-Blind, Randomized, Placebo-Controlled, Single-Dose Two-Period Crossover Study to Assess the Efficacy of KAI-1678 Administered by Subcutaneous Infusion in Subjects With Spinal Cord Injury
Brief Title: Safety and Efficacy Study of KAI-1678 to Treat Pain in Subjects With Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Collaborators: Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KAI-1678-004
Record Dates: First submitted 2010-04-16; First posted 2010-06-02 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
Keywords: Analgesics. Non-narcotic / therapeutic use; Spinal Cord Injuries; Pain; Pain measurement / drug effect; Pain postoperative / drug therapy
MeSH Terms: conditions — Spinal Cord Injuries; Pain; Pain, Postoperative | interventions — KAI-1678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1: Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- A2: KAI-1678 (Experimental): Experimental
  Interventions: Drug: KAI-1678

INTERVENTIONS:
Drug: Placebo — Placebo IV Infusion
  Arms: A1: Placebo
Drug: KAI-1678 — KAI-1678 IV Infusion
  Arms: A2: KAI-1678

SUMMARY:
The purpose of this study is to determine whether KAI-1678 is effective in the treatment of pain associated with spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury at least 1 year prior and nonprogressive ofr at least 6 months
* central neuropathic pain for at least 3 months or with relapses and remissions for at least 6 months
* pain score at least 4 on 11-point numerical rating scale (0-10)
* stable doses of analgesic medications for at least 1 month

Exclusion Criteria:

* history of chronic alcoholism or chronic substance abuse
* tolerance to opioid analgesics
* clinically significant abnormality on laboratory tests or ECG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The effect of KAI-1678 on mean change from baseline in pain intensity at 6 hours (PID 6). | 6 hours

SECONDARY OUTCOMES:
The effect of KAI-1678 on the proportion of subjects achieving at least a 1 point improvement in pain intensity at 6 hours | 6 hours
The effect of KAI-1678 on patient global impression of change | 6 hours
The effect of KAI-1678 on symptoms of neuropathic pain assessed by the Neuropathic Pain Scale (NPS) | 6 hours
The number of participants with adverse events as a measure of safety and tolerability of KAI-1678 | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals, Inc
Locations (1):
- Sydney, New South Wales, Australia